CLINICAL TRIAL: NCT06228001
Title: Holter of Movement in Patients With Amyotrophic Lateral Sclerosis.
Acronym: ActiALS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: SYSNAV (Industry)
Responsible Party: Principal Investigator, Laurent Servais, Professor, Centre Hospitalier Universitaire de Liege
Other Study IDs: ActiALS study
Record Dates: First submitted 2023-12-14; First posted 2024-01-29 (Actual); Last update posted 2025-05-19 (Actual); Status verified 2025-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Actimyo; Accelerometry; Daily living
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Actimyo — Actimyo is an innovative device intended to be used in a home-based environment. It is composed of two watch-like sensors, each containing a magneto-inertial sensors that record the linear acceleration, the angular velocity, the magnetic field of the movement in all directions.The two watches can be worn as wristwatch or placed near the ankle.

SUMMARY:
ActiALS is a multicentric academic study. Patients with amyotrophic lateral sclerosis (ALS) may be included on a voluntary basis. The investigators plan to include a group of approximately 30 patients with ALS.

The investigators have planned to assess patient every three months for a year. After each visit, participants will wear Actimyo for one month daily.

DETAILED DESCRIPTION:
On each visit, participants will undergo a clinical examination with MRC sum score and Ashworth scores.

Participants will perform few tests (6-minutes walk test (6MWT), dynamometric measure, electromyography, and will answer to some questionaires (dysphagia handicap scale, Revised Amyotrophic Lateral Sclerosis Functional Rating Scale).

Actimyo is an innovative device intended to be used in a home-based environment. It is composed of two watch-like sensors, each containing a magneto-inertial sensors that record the linear acceleration, the angular velocity, the magnetic field of the movement in all directions.The two watches can be worn as wristwatch or placed near the ankle.

ELIGIBILITY:
Inclusion Criteria:

* Clinically defined or probable diagnosis of ALS according to El Escorial criteria revised with Awaji's electro-diagnostic algorithm.
* Over 18 years old.
* Signed informed consent
* If patient on Riluzole, the dosage should be stable for 1 month and continued throughout the study period.

Exclusion Criteria:

* Patients with excessive cognitive disorders, limiting the understanding of task or with apparent communication difficulties hindering data collection.
* Any other previous or present pathology having an impact on motor function.
* Recent surgery or trauma (less than 6 months) in the upper or lower limbs.
* Prior neurological, endocrine, infectious, allergic, or chronic or acute inflammatory pathology in the three weeks preceding inclusion.
* Patients participating in an interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with amyotrophic lateral sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Difference in 95th centile of stride velocity between baseline and one year follow up- or last time point | 1 year
  95th centile of stride velocity obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter per second).
Difference in 50th centile of stride velocity between baseline and one year follow up- or last time point | 1 year
  50th centile of stride velocity obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter per second).
Difference in 95th centile of stride length between baseline and one year follow up- or last time point | 1 year
  95th centile of stride length obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter).
Difference in 50th centile of stride length between baseline and one year follow up- or last time point | 1 year
  50th centile of stride length obtained with a magneto-inertial sensor (Actimyo°) in real-life (meter).

SECONDARY OUTCOMES:
Upper limb function evolution in patient with ALS | 1 year
  Upper limb function assessed with a magneto-inertial sensor (Actimyo°) in real-life.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Delstanche, MD, Principal Investigator — Centre de référence des maladies neuromusculaire, Centre Hospitalier Régional de la Citadelle
Locations (3):
- Belgium (2):
  - Katholieke Universiteit Leuven, Leuven
  - Centre de référence des maladies neuromusculaire, Centre Hospitalier Régional de la Citadelle, Liège
- Galaa Military Medical Complex, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No